CLINICAL TRIAL: NCT06892717
Title: Caregiver Burden and Associated Factors in Parkinson's Disease
Brief Title: Caregiver Burden in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH16
Record Dates: First submitted 2025-03-08; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Primary caregivers of patients diagnosed with idiopathic Parkinson's disease will be included in the study. A total of 43 participants will be recruited. At the beginning of the study, demographic data and clinical characteristics of the patients, including disease stage, history of falls, presence of fractures, presence and severity of pain, comorbidities, and medication use, will be recorded.

Subsequently, caregivers' age, gender, occupation, relationship to the patient, caregiving duration, and their own comorbidities will be assessed. Sleep problems will be evaluated using the Insomnia Severity Index (ISI), while symptoms related to depression and anxiety will be assessed with the Hospital Anxiety and Depression Scale (HADS). Caregiver burden will be examined using the Zarit Caregiver Burden Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-80 years
* Diagnosed with Parkinson's disease, Hoehn and Yahr stage 2-5
* Requires assistance in daily activities
* Informal caregiver providing care (unpaid, typically a family member such as a spouse or child)
* Caregiver has sufficient proficiency in Turkish to understand and respond to the study questions

Exclusion Criteria:

* Presence of any additional neurodegenerative disease other than Parkinson's disease
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Advanced heart failure classified as New York Heart Association (NYHA) Class IV (symptoms at rest)
* Active cancer disease
* History of stroke causing limitations in daily life
* Immobility due to reasons other than Parkinson's disease

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of caregivers of patients diagnosed with Parkinson's disease, aged between 40-80 years, who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Zarit Caregiver Burden Scale | Baseline
  A scale used to assess the physical, emotional, and social burden of caregiving, with higher scores indicating greater caregiver burden. Score range: 0-88.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline
  A scale used to evaluate the severity of sleep problems in caregivers, with higher scores reflecting more severe insomnia. Score range: 0-28.
Hospital Anxiety and Depression Scale (HADS)- Anxiety score | Baseline
  A tool used to assess symptoms of anxiety in caregivers. Higher scores indicate more severe anxiety. Score range: 0-21.
Hoehn and Yahr Scale | Baseline
  A classification system used to determine the disease stage of Parkinson's disease, with higher stages indicating more severe disease progression. Score range: 1-5.
Visual Analog Scale (VAS) | Baseline
  A linear scale used to assess pain severity, where higher scores indicate more severe pain. Score range: 0-10.
Hospital Anxiety and Depression Scale (HADS)- Depression score | Baseline
  A tool used to assess symptoms of depression in caregivers. Higher scores indicate more severe depressive symptoms. Score range: 0-21.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No